CLINICAL TRIAL: NCT01629082
Title: Clofarabine Followed by Lenalidomide for Treatment of High Risk Myelodysplastic Syndromes and Acute Myeloid Leukemia
Brief Title: Clofarabine Followed By Lenalidomide for High-Risk Myelodysplastic Syndromes and Acute Myeloid Leukemia
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Collaborators: Celgene Corporation (Industry)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 120146; 12-H-0146
Record Dates: First submitted 2012-06-22; First posted 2012-06-27 (Estimated); Last update posted 2019-12-17 (Actual); Status verified 2018-06-27

CONDITIONS: Myeldysplastic Syndrome (MDS); Chronic Myelomonocytic Leukemia; Bone Marrow Diseases; Neutropenia; Acute Myeloid Leukemia (AML)
Keywords: Myelodysplastic Syndromes; Acute Myeloid Leukemia (AML); Chronic Myelomonocytic Leukemia (CMML)
MeSH Terms: conditions — Leukemia, Myelomonocytic, Chronic; Bone Marrow Diseases; Neutropenia; Leukemia, Myeloid, Acute; Myelodysplastic Syndromes | interventions — Clofarabine; Lenalidomide

INTERVENTIONS:
Drug: Clofarabine
Drug: Lenalidomide

SUMMARY:
Background:

* Several types of blood cancer are associated with poor outcomes including high-risk myelodysplastic syndromes (MDS), chronic myelomonocytic leukemia (CMML) and acute myelogenous leukemia (AML). Many people with MDS, CMML, and AML are not candidates for standard treatments. New types of treatment are needed for these cancers.
* Clofarabine and lenalidomide are anticancer drugs. The first damages cancer cells in the body. The second can alter blood supply to abnormal cells or affect how the immune system attacks these cells. These drugs have been previously tested as treatments for MDS and leukemia. However, they have not been tried as a combination for MDS, CMML, and AML. Researchers want to see if these drugs are safe and effective for these types of cancer.

Objectives:

- To test the safety and effectiveness of clofarabine and lenalidomide for people with high-risk MDS, CMML, and AML.

Eligibility:

* Individuals at least 18 years of age who have high-risk MDS, CMML, and AML.
* Participants must not be candidates for standard treatments.

Design:

* Participants will be screened with a physical exam and medical history. Blood and bone marrow samples will be collected.
* Participants will have 5 days of treatment with clofarabine. It will be given through a vein during an inpatient hospital stay. If there are no serious side effects after the infusion, participants will continue treatment as outpatients.
* After 28 days, participants will have a bone marrow biopsy to check their response to treatment.
* After the biopsy, participants will start lenalidomide treatment. Half of the participants will take the drug for 28 days (one treatment cycle). The other half will take it for 56 days (two cycles). More blood tests and biopsies will be used to monitor treatment.
* If there are no serious side effects and the disease does not become worse, participants may keep taking lenalidomide at lower doses for up to 12 more cycles.

DETAILED DESCRIPTION:
High risk myelodysplastic syndromes (MDS), chronic myelomonocytic leukemia (CMML) and acute myelogenous leukemia (AML) are hetereogeneous myeloid malignancies that are associated with a poor prognosis. Due to advanced age and medical comorbidities, the majority of MDS, CMML, and AML patients are not candidates for potentially curative standard treatments such as allogeneic stem cell transplantation (SCT) or intensive chemotherapy (ICT). New therapeutic approaches that improve response rates, have lesser toxicity, and extend survival are clearly needed for high risk MDS and AML patients.

Clofarabine is a myelosuppressive, second generation purine nucleoside analogue which has shown meaningful efficacy at variable dosing levels for high risk MDS and AML patients with a favorable toxicity profile compared to intensive chemotherapy. Lenalidomide is an oral structural analogue of thalidomide with a complex mechanism of action including immunomodulatory, anti-angiogenic, and direct cytotoxic effects which is a well-established treatment for MDS and has shown agent single efficacy at higher doses for AML. Lenalidomide s therapeutic benefit in AML has been the greatest in patients with low presenting total leukocyte and circulating blast counts. We hypothesize that the initial cytoreductive effects of clofarabine may augment the effectiveness of subsequent lenalidomide therapy and create a favorable immunologic milieu for patients eligible for lenalidomide maintenance therapy. This open-label, single institution phase I trial will evaluate a sequential combination of IV clofarabine with oral lenalidomide for the treatment of high risk MDS, CMML, and AML. Subjects will receive a single course of IV clofarabine (5 milligrams per metered square per day times 5) for cytoreduction. This will be followed by oral lenalidomide consolidation with dose escalation from 25 mg daily for 21/28 days for 1 cycle in the first cohort up to 50 mg daily for 28/28 days for 2 cycles in the fourth cohort. In the absence of dose limiting toxicity or disease progression, Subjects will receive lenalidomide maintenance, starting at a dose of 10 mg daily in 28 day cycles, with dose adjustments, for up to 12 cycles.

The overall objective is to determine the safety of sequential therapy with clofarabine and lenalidomide in subjects with high risk MDS, CMML, and AML. The primary study endpoint will be the toxicity profile of this novel treatment combination in each cohort. Secondary endpoints will include characterization of response and duration, overall survival, and the feasibility of maintenance lenalidomide therapy for responding subjects.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Age greater than or equal to 18 years old
* Unequivocal diagnosis of MDS (including chronic myelomonocytic leukemia- CMML) according to WHO criteria with IPSS risk categorization for MDS subjects of intermediate-2 to high confirmed by bone marrow evaluation within 30 days prior to study enrollment

OR

Unequivocal diagnosis of AML according to WHO criteria to include secondary and relapsed or refractory disease confirmed by bone marrow evaluation within 30 days prior to study enrollment

* ECOG Performance Status less than or equal to 2
* Must have failed at least one prior therapy before study enrollment
* Ability to comprehend the investigational nature of the study and provide informed consent
* All study participants must be registered into the mandatory RevAssistRevlimid REMS program, and be willing and able to comply with the requirements of RevAssistRevlimid REMS .
* Females of childbearing potential (FCBP) must have a negative serum or urine pregnancy test with a sensitivity of at least 50 mIU/mL within 10 14 days and again within 24 hours prior to prescribing lenalidomide for Cycle 1 (prescriptions must be filled within 7 days as required by RevAssistRevlimid REMS ) and must either commit to continued abstinence from heterosexual intercourse or begin TWO acceptable methods of birth control, one highly effective method and one additional effective method AT THE SAME TIME, at least 28 days before she starts taking lenalidomide. FCBP must also agree to ongoing pregnancy testing. Females of reproductive potential must adhere to the scheduled pregnancy testing as required in the Revlimid REMSTM program. Men must agree to use a latex condom during sexual contact with a FCBP even if they have had a successful vasectomy.

EXCLUSION CRITERIA:

* Prior Allogeneic Stem Cell Transplant
* Diagnosis of acute promyelocytic leukemia
* Diagnosis of atypical chronic myeloid leukemia BCR-ABL1 negative, juvenile myelomonocytic leukemia, yelodysplastic/myeloproliferative neoplasm unclassifiable)
* Prior therapy with clofarabine at any dose
* Prior therapy with lenalidomide at doses greater than or equal to 25 milligrams daily
* Clinically significant active infection not responding adequately to therapy
* HIV Positive
* Uncontrolled concurrent hepatic, renal, cardiac, pulmonary, neurologic, infectious, or metabolic disease of such severity, which in the opinion of the PI, would preclude the subjects s ability to tolerate protocol therapy
* Ejection fraction less than 40% by Echocardiogram or MUGA
* Calculated creatinine clearance less 60 milliliters per minute
* Serum bilirubin greater than 1.5 times upper limit of normal
* Aspartate aminotransferase (AST) or Alanine aminotransferase (ALT) greater than 3 times upper limit normal
* Decreased oxygen saturation at rest (e.g. pulse oximeter less than 88% or PaO2 less than or equal to 55 millimeters of mercury)
* Patients with any condition that prevents their ability to swallow and retain lenalidomide tablets
* Severe psychiatric illness or complex social situations that would limit the patient s ability to tolerate and/or comply with study requirements
* Current pregnancy or breastfeeding

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2012-06-06; Primary Completion 2015-10-27 (Actual); Study Completion 2018-06-27 (Actual)

PRIMARY OUTCOMES:
Identification of the maximum tolerated dose.

SECONDARY OUTCOMES:
Overall Survival
Characterization of response rate and duration
Feasibility of lenalidomide maintenance therapy

CONTACTS AND LOCATIONS:
Overall Officials: Sawa Ito, M.D., Principal Investigator — National Heart, Lung, and Blood Institute (NHLBI)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Garcia-Manero G, Fenaux P. Hypomethylating agents and other novel strategies in myelodysplastic syndromes. J Clin Oncol. 2011 Feb 10;29(5):516-23. doi: 10.1200/JCO.2010.31.0854. Epub 2011 Jan 10. PMID 21220589
- [Background] Aul C, Gattermann N, Schneider W. Age-related incidence and other epidemiological aspects of myelodysplastic syndromes. Br J Haematol. 1992 Oct;82(2):358-67. doi: 10.1111/j.1365-2141.1992.tb06430.x. PMID 1419819
- [Background] Rollison DE, Howlader N, Smith MT, Strom SS, Merritt WD, Ries LA, Edwards BK, List AF. Epidemiology of myelodysplastic syndromes and chronic myeloproliferative disorders in the United States, 2001-2004, using data from the NAACCR and SEER programs. Blood. 2008 Jul 1;112(1):45-52. doi: 10.1182/blood-2008-01-134858. Epub 2008 Apr 28. PMID 18443215